CLINICAL TRIAL: NCT05457491
Title: Novel Antiaging Regenerative Skin Care Regimen Containing Human Platelet Extract (HPE)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator discretion
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Saranya P. Wyles, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-008529
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Skin Aging
MeSH Terms: interventions — Cosmetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Human platelet extract (HPE) (Experimental): Subjects will follow a standardized twice daily skin care regimen of applying morning and night. Morning skin care routine includes Vanicream Gentle Facial Cleanser, human platelet extract, and EltaMD UV Daily Broad-Spectrum SPF 40, or Vanicream Lite Lotion. Evening skin care routine includes Vanicream Gentle Facial cleanser, human platelet extract, and EltaMD PM Therapy Facial Moisturizer or Vanicream Lite Lotion
  Interventions: Biological: Human platelet extract (cosmetic product); Other: Vanicream Gentle Facial Cleanser; Other: EltaMD UV Daily Broad-Spectrum SPF 40; Other: EltaMD PM Therapy Facial Moisturizer; Other: Vanicream Lite Lotion

INTERVENTIONS:
Biological: Human platelet extract (cosmetic product) — A leukocyte depleted allogeneic product derived from human U.S. sourced pooled apheresed platelets (derived from screened healthy donors). Applied to face twice daily for 12 weeks.
Other: Vanicream Gentle Facial Cleanser — A mild cleanser specifically formulated for daily facial use. Applied to face twice daily for 12 weeks
Other: EltaMD UV Daily Broad-Spectrum SPF 40 — A daily moisturizer with a lightweight formula that provides broad-spectrum sunscreen protection. EltaMD UV Daily Broad-Spectrum SPF 40 provides powerful protection against the sun's harmful UV rays, as it hydrates and is gentle enough for post-procedure skin. Powered by hyaluronic acid, this face sunscreen plumps the skin with lightweight moisture, while micronized zinc and octinoxate shield skin from UVA/UVB rays to prevent the visible signs of environmentally caused aging. Applied to face once daily for 12 weeks.
Other: EltaMD PM Therapy Facial Moisturizer — A fortifying face moisturizer to repair elasticity and vitality. EltaMD PM Therapy Facial Moisturizer restores youthfulness while strengthening the skin's natural moisture barrier. Niacinamide blends with antioxidants to boost the skin color and tone, as it speeds up the skin's repair processes. Rice protein peptides aid in encouraging cell growth, promoting collagen formation and improving elasticity. Applied to face once daily for 12 weeks.
Other: Vanicream Lite Lotion — Lotion to restore and maintain a normal moisture level. Applied to face twice daily for 12 weeks.

SUMMARY:
The Researchers are trying to study a cosmetic skin care product called human platelet extract (HPE) to see if it can be used as a possible treatment for skin anti-aging and skin rejuvenation. They are trying find out the safety and tolerability of topical HPE after multiple doses of topical administration

ELIGIBILITY:
Inclusion Criteria:

* Persons of childbearing potential must have a negative pregnancy test prior to receiving the study product and will agree to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 2 years until discontinuation of treatment. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study product to confirm negative results. If the urine pregnancy test is positive, the study product will not be administered, and the result will be confirmed by a serum pregnancy test. Urine pregnancy tests will be performed by qualified personnel using kit. Persons becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any Serious Adverse Events (SAE) associated with pregnancy will be recorded.
* All skin phototypes ≥ grade I of Fitzpatrick's classification.
* Mild-to-moderate global face wrinkles and mild-to-moderate global fine lines based on a modified Griffiths' 10-point scale [3].
* Fully understanding of the requirements of the study and willingness to comply with the treatment plan, including laboratory tests, diagnostic imaging, and follow-up visits and assessments.
* Volunteer willingness to discontinue any other anti-aging topical or parenteral treatments for the duration of the study.
* Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related treatment.
* Can provide written informed consent to being photographed for purposes of treatment for medical, scientific purposes.

Exclusion Criteria:

* Pregnant or nursing, or planning on becoming pregnant during the study period
* Subjects who have had an antiaging or aesthetic treatment prior to the study: Botox or Botox-like products, peelings, plastic surgery, resurfacing with Laser, Intense pulsed light (IPL) therapy, threats, radiofrequency treatments, hyaluronic acid treatment, Plasma-Rich Platelets treatment, or any other specific treatments prone to change the skin aspect during the last 6 months
* Individuals with a history of any dermatological disease or condition, including but not limited to active atopic dermatitis, psoriasis, eczema, active seasonal allergies, collagen diseases, or skin cancer involving the treated sites within the past 6 months
* Cutaneous marks on the experimental area which could interfere with the assessment of skin reactions (pigmentation problems, scar elements, over-developed pilosity, ephelides, and nevi in too great quantity, sunburn, beauty spots, freckles, etc.)
* Participants with asymmetric photodamage on dorsal hands due to environmental exposures (i.e., golfing) and/or other skin lesions including burns or scars resulting in significant skin surface variability between dorsal hands
* Eczematous reaction still visible, scar, or pigmentary sequelae of previous tests on the experimental area
* Allergy to colophony or nickel.
* Allergy or reactivity to drugs, food or cosmetic products previously observed, including perfumes or cologne products.
* Skin hyper-reactivity.
* Forecast of intensive sun, tanning bed use or UV phototherapy during the test period.
* Treatment with prescription-strength Vitamin A acid or its derivatives within 3 months before the beginning of the study.
* Treatment with topical steroids on the experimental area within 16 days before the study.

Study constraints:

* No application of products on the experimental area (except the suggested ones), particularly any anti-aging cosmetic products except for sunscreen.
* No change in hygiene habits
* No application of any cosmetic moisturizing products on the face or any makeup on face and lips, on the day of study evaluations
* No change in the way of life or in the physical activity
* No change in dietary activities, or any treatment that significantly impacts body weight
* No exfoliating treatment on the experimental areas
* Description of any treatment undertaken during the study and all eventual deviations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saranya P Wyles, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Platelet Extract (HPE): Subjects followed a standardized twice daily skin care regimen of applying morning and night for 12 weeks. Morning included Vanicream Gentle Facial Cleanser, human platelet extract, and EltaMD UV Daily Broad-Spectrum SPF 40, or Vanicream Lite Lotion. Evening skin care routine included Vanicream Gentle Facial cleanser, human platelet extract, and EltaMD PM Therapy Facial Moisturizer or Vanicream Lite Lotion.
  Human platelet extract is a leukocyte depleted allogeneic product derived from human U.S. sourced pooled apheresed platelets (derived from screened healthy donors. Vanicream Gentle Facial Cleanser is a mild cleanser specifically formulated for daily facial use. EltaMD UV Daily Broad-Spectrum SPF 40 is a daily moisturizer with a lightweight formula that provides broad-spectrum sunscreen protection. EltaMD PM Therapy Facial Moisturizer is a fortifying face moisturizer to repair elasticity and vitality. Vanicream Lite Lotion is a lotion to restore and maintain a normal moisture level.
Period: Overall Study
Arm/Group | Human Platelet Extract (HPE)
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Redness Area
Description: The percentage of participants to experience at least 50% improvement in redness area over baseline. As measured by photodocumentation with the VISIA-CR Generation 5 3D PRIMOS using RBX technology. Redness pixel variation and the cross polarized image were transformed into red images that correlated with hemoglobin absorption/distribution.
Time Frame: baseline, 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 55
percentage of participants | 42

2. Primary Outcome: Change Brown Spot Area
Description: Photodocumentation with the VISIA-CR Generation 5 3D PRIMOS to assess overall variation in color values specifically pixel variation across defined cosmetic subunits and how rapidly those colors change spatially within it, producing a score from 0 to 1, where 0 is less melanin or brown color and 1 is more melanin or brown color. Lower scores reflect better outcomes.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 55
pixels
  Baseline | 0.097 (0.030)
  6 weeks | 0.093 (0.031)

3. Primary Outcome: Change in Luminosity
Description: Luminosity (color intensity) is the measure of the light reflected from the skin surface. Photodocumentation with the VISIA-CR Generation 5 3D PRIMOS to assess overall variation in color values specifically pixel variation across defined cosmetic subunits and how rapidly those colors change spatially within it. Lower values reflect dull and/or uneven skin tones. Higher values reflect radiant and/or even-appearing skin tones.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 55
pixels
  Baseline | 60.29 (5.49)
  6 weeks | 63.19 (5.24)

4. Primary Outcome: Change in Color Evenness
Description: Photodocumentation with the VISIA-CR Generation 5 3D PRIMOS to assess overall variation in color values specifically pixel variation across defined cosmetic subunits and how rapidly those colors change spatially within it, producing a score from 0 to 1, where 0 is dull and/or uneven skin tone and 1 is radiant and/or even-appearing skin tone. Higher scores reflect better outcomes.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 55
pixels
  Baseline | 0.51 (0.07)
  6 weeks | 0.54 (0.07)

5. Primary Outcome: Change in Wrinkles Area
Description: Photodocumentation with the VISIA-CR Generation 5 3D PRIMOS to assess forehead wrinkles using 3D fringe projection which evaluates static wrinkles and measures the difference in fractional area change
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 55
pixels
  Baseline | 0.08 (0.03)
  6 weeks | 0.09 (0.03)

6. Secondary Outcome: Cosmetic Skin Improvement
Description: Change measured by the self reported Global Aesthetic Improvement Assessment where subjects grade/rate their improvement as Exceptional/very much improved, Moderate/much improved, Slight, No change or Worse.
Time Frame: 12 weeks
Population: Terminated study. Data was not collected nor analyzed
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 0

7. Secondary Outcome: Satisfaction With Topical Cosmetic Treatment
Description: Number of subjects to self report satisfied or very satisfied with the treatment on the Modified Cosmetic Improvement questionnaire.
Time Frame: 12 weeks
Population: Data was not collected nor analyzed
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 0

8. Secondary Outcome: Recommendation of Topical Cosmetic Treatment
Description: Number of subjects to self report they would recommend the treatment to a friend on the Modified Cosmetic Improvement questionnaire.
Time Frame: 12 weeks
Population: Terminated study. Data was not collected nor analyzed
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 0

9. Secondary Outcome: Likelihood of Continuing Topical Cosmetic Treatment
Description: The number of subjects to self report they are very likely to continue treatment on the Modified Cosmetic Improvement questionnaire.
Time Frame: 6 weeks
Population: One subject did not complete the questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 55
Participants | 54

10. Secondary Outcome: Topical Cosmetic Treatment on Self-esteem
Description: Number of subjects to self report how the cosmetic treatment affected self-esteem positively or negatively on the Modified Cosmetic Improvement questionnaire.
Time Frame: 12 weeks
Population: Terminated study. Data was not collected nor analyzed
Arm/Group | Human Platelet Extract (HPE)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for all subjects from baseline to end of study, approximately 12 weeks
Arm/Group | Human Platelet Extract (HPE)
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 9/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Human Platelet Extract (HPE) (N=56)
Dry Skin (Skin and subcutaneous tissue disorders) | 9

LIMITATIONS AND CAVEATS:
Study was terminated early per Principal Investigator

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT05457491/Prot_SAP_000.pdf